CLINICAL TRIAL: NCT01805336
Title: Assessment of Attentional and Executive Disorders in Multiple Sclerosis Using Techniques of Virtual Reality
Acronym: SEPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2012-A000000166-37; 12-027 (Other: CaenUH)
Record Dates: First submitted 2013-02-26; First posted 2013-03-06 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2020-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Relapsing-Remitting MS; cognitive impairment; virtual reality
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Other): Inclusion : cognitive complaint,fatigue, anxiety an depression questionnaires.
  Assessment 1 : attentional function by traditional tests + executive function by virtual reality tests.
  One week later, Assessment 2 : attentional function by virtual reality tests + executive function by traditional tests.
  Interventions: Other: Assessment of attentional functions by traditional tests; Other: Assessment of attentional functions by virtual reality tests; Other: Assessment of executive functions by traditional tests; Other: Assessment of executive functions by virtual reality test; Other: Evaluation of cognitive complaint, fatigue, anxiety and depression
- Arm B (Other): Inclusion : cognitive complaint,fatigue, anxiety an depression questionnaires.
  Assessment 1 : attentional function by virtual reality tests + executive function by traditional tests.
  One week later, Assessment 2 : attentional function by traditional tests + executive function by virtual reality tests.
  Interventions: Other: Assessment of attentional functions by traditional tests; Other: Assessment of attentional functions by virtual reality tests; Other: Assessment of executive functions by traditional tests; Other: Assessment of executive functions by virtual reality test; Other: Evaluation of cognitive complaint, fatigue, anxiety and depression

INTERVENTIONS:
Other: Assessment of attentional functions by traditional tests — For assessment of attentional functions, traditional tests include : Symbol Digit Modalities Test (SDMT), Test d'Evaluation de l'Attention (TEA), Attentional Network Test (ANT).
Other: Assessment of attentional functions by virtual reality tests — For assessment of attentional functions, virtual reality tests include : Monotonous task of driving on motorways, Task of city driving with accident scenarios, Monotonous driving task with divided attention test ; all tests realized on a driving simulator.
Other: Assessment of executive functions by traditional tests — For assessment of executive functions, traditional tests include : Wisconsin Card Sorting Test (WCST), Task verbal fluencies, Sequence Numbers Letters subtest of the Wechsler Adult Intelligence Scale (WAIS) III, Commissions.
Other: Assessment of executive functions by virtual reality test — For assessment of executive functions, virtual reality test include : VAP-S.
Other: Evaluation of cognitive complaint, fatigue, anxiety and depression — The following questionnaires will be completed by the participant at the inclusion visit : cognitive complaint RBN-SEP questionnaire to assess cognitive complaint, EMIF-SEP to assess fatigue, STAI (State Trait Anxiety Inventory) to assess anxiety and MADRS to assess depression.

SUMMARY:
Since many years cognitive disorders are a main topic of clinical research in Multiple Sclerosis (MS) as there could be observed early on in the disease and could induce with time in patients significant socio-professional burden. Today assessment of cognitive dysfunction in MS is still based on traditional pencil-paper task tests which are not able to give a true representation of functional burden observed in patients in real life situations. The development of new tools close to these "life situations", i.e. more ecological, are needed to better assess and take in charge cognitive impairment in MS patients. One way to reach this goal is Virtual Reality (VR). VR offers a new human-computer interface paradigm that simulates a realistic 3D environment where the user become immersed and interacts with it. These last ten years VR has known a rapid development in the health domain and has been applied with success to motor rehabilitation, psychiatry and neuropsychology. In this last domain, virtual environment (VE) reproducing activities of daily living have been used to evaluate executive and memory functions as well as attentional or visuospatial processes. Among main VE developed, driving assessment system, navigation skills, cooking behaviors, virtual supermarket have shown better sensitivity to detect functional consequences of cognitive impairment in various neurological and psychiatric disorders than traditional evaluations. In Caen University Hospital, investigators used VE driving system and developed the use of the Virtual Action Planning in a supermarket (VAP-S ; Klinger et al 2004) where a user move to select and buy groceries and other things inside an interactive virtual supermarket using a shopping cart. In a preliminary study investigators have used this virtual interactive tool to evaluate executive functioning in small group of Parkinson's disease and MS patients. Analysis of initial data shows the feasibility of the VAP-S for use with these two kinds of diseases. According to these results investigators planned a new study in Relapsing-Remitting(RR)- MS patients where they compare the use of VE (driving system and the VAP-S) to traditional attentional and executive evaluation for estimate their respective sensitivity to detect cognitive/functional impairment in MS patients. Investigators hope to shown that VR will demonstrate its interest to assess cognitive functions in MS and to develop cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients only :

  * Diagnosis of RR-MS in accordance with the Polman et al. criteria (2011)
  * Expanded Disability Status Scale (EDSS) < 6
  * Any disease duration
* Patients and healthy subjects :

  * Men and women
  * Ages 30-60 years inclusive
  * Score of > 130 on the Mattis Dementia Rating Scale (DRS)
  * Score of < 15 on the Montgomery and Asberg Depression Rating Scale (MADRS)
  * French native language
  * Licensed drivers (> 2 years)
  * Experienced drivers (> 5000 km / year)
  * Normal or corrected visual acuity greater than or equal to 6/10
  * Sign informed consent

Exclusion Criteria:

* Patients only :

  * Any relapse or corticosteroids therapy within 30 days
  * Under guardianship
* Patients and healthy subjects

  * Other neurological, psychiatric or developmental disease
  * Serious systemic disease
  * Sequelae of brain injury
  * Antidepressants or anxiolytics treatment within 4 weeks
  * Treatment known to interfere with cognition (e.g. psychostimulant) within 3 months
  * Alcohol > 28 units / week
  * Addiction
  * Cognitive assessment within a year (including all or part of the assessment proposed in this study)
  * Sensory or motor failure incompatible with study tasks

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Scores for traditional tests | 2 visits over 1 week
  For each test, scores will be compared between patients and healthy subjects.
Scores for virtual reality tests | 2 visits over 1 week
  For each test, scores will be compared between patients and healthy subjects.
Correlation between traditional and virtual reality tests | 2 visits over 1 week
  Links between scores for traditional tests and scores for virtual reality tests will assessed by calculating Pearson or Spearman correlation coefficents, among all participants.
Z-scores for traditional and virtual reality tests | 2 visits over 1 week
  For each patient and each score, z-score will be calculated. For traditional and virtual reality tests for which a correlation will be observed, the z-scores will be compared.

SECONDARY OUTCOMES:
Score for cognitive complaint questionnaire | Inclusion visit
  Correlation coefficients will be calculated between scores for cognitive complaint questionnaire and scores for virtual reality tests, among all participants.
Scores for fatigue, anxiety and depression questionnaires | inclusion visit
  Correlation coefficients will be calculated between scores for fatigue, anxiety and depression questionnaires and scores for traditional and virtual reality tests, among all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Defer, Professor, Principal Investigator — University Hospital, Caen
Locations (2):
- France (2):
  - Department of Neurologie, Caen Hospital University, Caen, Basse-Normandie
  - Inserm Unit 1075 Comete, Caen Hospital University, Caen, Basse-Normandie